CLINICAL TRIAL: NCT04499963
Title: An Open-label, Single-center, 6-month Trial of Theracurmin for Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Trial of Theracurmin for Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Richard Bedlack, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Richard Bedlack, M.D., Ph.D., Professor of Neurology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103700
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: This will be a 6-month, widely inclusive, largely remote/virtual, single-center, open-label pilot trial utilizing a historical control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open Label Arm (Experimental): The intervention is twice daily dosage of Theracurmin 90 mg capsules. This same dose was used in a successful trial of patients with mild cognitive impairment. Theracurmin HP capsules containing 90 mg curcumin each that will be taken as one capsule twice daily for 6 months. Each capsule contains 300 mg Theracurmin enhanced bioavailable water-dispersible turmeric rhizome complex providing 30% curcumin (90 mg). The content of Theracurmin HP has been independently certified by NSF International under NSF/ANSI 173.
  Interventions: Drug: Theracurmin HP
- Healthy Control Arm (No Intervention): We will seek to enroll 50 healthy control participants. We will attempt to enroll one control subject from each enrolled primary participant's home, preferably a spouse or partner of similar age if possible. We plan to use this data to compare the microbiome of control participants to that of the ALS participants at baseline, week 4 and month 6. We will not conduct further follow-up or collect additional samples with the control subjects.

INTERVENTIONS:
Drug: Theracurmin HP — The intervention is based on the twice daily dosage of Theracurmin 90 mg capsules used in a trial of patients with mild cognitive impairment
  Arms: Open Label Arm

SUMMARY:
This will be a 6-month, widely inclusive, virtual, single-center, open-label pilot trial utilizing a historical control group.

DETAILED DESCRIPTION:
This will be a 6-month, widely inclusive, virtual, single-center, open-label pilot trial utilizing a historical control group. Following informed consent and screening, participants with ALS will take Theracurmin 1 capsule (90mg) twice daily for 6-months. Treatment with the Theracurmin and all study outcome measures and labs are being performed exclusively for research purposes. Collected data includes saliva and stool microbiome sampling, adverse events, concomitant medications, weight and height, Theracurmin treatment evaluations, and Thrive Questionnaires. Participants will be asked to register on the website Patientslikeme.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years.
* Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria.
* Patient is able to understand and express informed consent (in the opinion of the site investigator).
* Patient has access to the Internet on a desktop computer, laptop, or tablet and has a working email address.
* Patient or caregiver is willing and able to use a computer and enter data on a secure website.
* Patient is able to read and write English.
* Patient is expected to survive for the duration of the trial.
* Women must not be pregnant (will have evidence of a negative pregnancy test obtained by local physician within past 7 days or be post-menopausal)
* Women must not be able to become pregnant (e.g., post-menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and three months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal contraception, for example patch or contraceptive ring), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.

Exclusion Criteria:

* Patient is taking other experimental treatments for ALS (those that are part of an active research study).
* Prior side effects from curcumin or turmeric containing products
* Patient has a medical or psychiatric illness that could in the investigator's opinion interfere with the patient's ability to participate in this study.
* Pregnant women or women currently breastfeeding.
* Life expectancy shorter than the duration of the trial.
* Taking an antiplatelet agent or anticoagulant (due to the theoretically increased risk of bleeding from curcumin products).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bedlack, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited through the Duke ALS Clinic over a 16 month period.
Pre-assignment Details: Patients with ALS who met inclusion criteria were enrolled into the Open Label Arm. The healthy control arm was for people without ALS who came from the same household as the patients.
Period: Overall Study
Arm/Group | Open Label Arm | Healthy Control Arm
Started | 50 | 50
Completed | 35 | 50
Not Completed | 15 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Death | 3 | 0
Not completed — Lack of Efficacy | 7 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics not collected on the healthy control arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label Arm | Healthy Control Arm | Total
Number analyzed (Participants) | 50 | 0 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.96 (11.46) |  | 60.96 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 |  | 19
  Male | 31 |  | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 3 |  | 3
  White | 43 |  | 43
  More than one race | 0 |  | 0
  Unknown or Not Reported | 3 |  | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 |  | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in ALSFRS-R Slope
Description: The ALSFRS-R (ALS Functional Rating Scale-Revised) will be determined at all video/telephone visits. ALSFRS-R is a quickly administered (five minute) ordinal rating scale (ratings 0-4) used to determine patients' assessments of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS. Change in ALSFRS-R scores correlate with change in strength over time, and it is closely associated with quality of life measures and predicted survival. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0=worst and 48=best.
Time Frame: Starting at week 4 and then once every 30 days for 6 months
Population: Participants with ALSFRS-R scores available.
Measure: Mean (Standard Deviation); unit: ALSFRS-R points per week
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 48 | 44
ALSFRS-R points per week | 0.229 (0.274) | 0.224 (0.194)
Statistical Analysis 1: Comparison: Open Label Arm; We compared he ALSFRS-R slope (not the actual score) of the patients in our open label treatment versus the historical controls; Test type: Superiority; p = 0.984, t-test, 2 sided

2. Secondary Outcome: Number of Participants With ALS Reversal
Description: Number of participants who have an ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised) score that improves by 4 points or more over 6 months. The ALSFRS-R is used to determine patients' assessments of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS. Change in ALSFRS-R scores correlate with change in strength over time, and it is closely associated with quality of life measures and predicted survival. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0=worst and 48=best.
Time Frame: Month 6
Population: Two open label arm participants withdrew consent after enrollment. Data not collected on the healthy control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 48 | 0
Participants | 0 |

3. Secondary Outcome: Total Number of Adverse Events as Measured by Patient Reporting
Description: Adverse and serious adverse events will be recorded throughout the study.
Time Frame: up to 6 months
Population: Two open label arm participants withdrew consent after enrollment. Data not collected on the healthy control arm.
Measure: Number; unit: adverse events
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 48 | 0
adverse events | 25 |

4. Secondary Outcome: Enrollment Rate
Description: The number of participants enrolled divided by the number of months it took to enroll them.
Time Frame: up to 6 months
Population: Data not collected on the healthy control arm.
Measure: Number; unit: participants per month
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 50 | 0
participants per month | 3.1 |

5. Secondary Outcome: Retention as Measured by the Number of Participants Who Completed the 6 Month Study Visit
Description: The percentage of enrolled participants who completed the 6 month study visit.
Time Frame: month 6
Population: Data not collected on the healthy control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 50 | 0
Participants | 35 |

6. Secondary Outcome: Shannon Diversity Index of the Oral Microbiome
Description: Comparing the changes in the saliva microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. Data will be compared within subjects with ALS to assess possible changes over the length of the study and identify microbial correlates of disease progression. The Shannon diversity index takes into account the number of species living in a habitat (richness) and their relative abundance (evenness). The minimum value is 0, which indicates no diversity (only one species is found). There is no upper limit to the index; the maximum value occurs when all species have the same number of individuals. Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: Shannon diversity index
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 45 | 42
Number analyzed (samples) | 117 | 107
Shannon diversity index
  Baseline: number analyzed (samples) | 45 | 42
  Baseline | 4.7 [1.5 to 6.2] | 4.7 [3.3 to 6.1]
  Post-treatment (months 1 and 6 combined): number analyzed (Participants) | 42 | 42
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 65
  Post-treatment (months 1 and 6 combined) | 4.7 [2.0 to 6.1] | 4.7 [2.8 to 6.5]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.05, Kruskal-Wallis

7. Secondary Outcome: Faith's Phylogenetic Diversity of the Oral Microbiome
Description: Comparing the changes in the saliva microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. Data will be compared within subjects with ALS to assess possible changes over the length of the study and identify microbial correlates of disease progression. Phylogenetic diversity (PD) is a measure of biodiversity, based on phylogeny (the tree of life). PD is defined as equal to the sum of the lengths of all the branches on the tree that span the members of the set. The branch lengths on the tree count the relative number of new features arising along that part of the tree. Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, and month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: units of PD
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 45 | 42
Number analyzed (samples) | 117 | 107
units of PD
  Baseline: number analyzed (samples) | 45 | 42
  Baseline | 13.5 [7.6 to 17.7] | 12.8 [8.6 to 17.3]
  Post-treatment (months 1 and 6 combined): number analyzed (Participants) | 42 | 42
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 65
  Post-treatment (months 1 and 6 combined) | 13.2 [8.3 to 19.3] | 12.7 [8.3 to 18.4]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.5, Kruskal-Wallis — Alpha Diversity

8. Secondary Outcome: Observed Features (Amplicon Sequence Variants, ASV) of the Oral Microbiome
Description: Comparing the changes in the saliva microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. Data will be compared within subjects with ALS to assess possible changes over the length of the study and identify microbial correlates of disease progression. An amplicon sequence variant (ASV) is any one of the inferred single DNA sequences recovered from a high-throughput analysis of marker genes. Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: ASVs
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 45 | 42
Number analyzed (samples) | 117 | 107
ASVs
  Baseline: number analyzed (samples) | 45 | 42
  Baseline | 121.4 [33.0 to 227.0] | 114.4 [43.0 to 226.0]
  Post-treatment (months 1 and 6 combined): number analyzed (Participants) | 42 | 42
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 65
  Post-treatment (months 1 and 6 combined) | 115.1 [40.0 to 209.0] | 110.6 [35.0 to 225.0]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.05, Kruskal-Wallis

9. Secondary Outcome: Pielou's Evenness Index of the Oral Microbiome
Description: Comparing the changes in the saliva microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. Data will be compared within subjects with ALS to assess possible changes over the length of the study and identify microbial correlates of disease progression. Pielou's evenness is an index that measures diversity along with species richness. While species richness is the number of different species in a given area, evenness is the count of individuals of each species in an area. A calculated value of Pielou's evenness ranges from 0 (no evenness) to 1 (complete evenness). Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: Pielou's evenness index
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 45 | 42
Number analyzed (samples) | 117 | 107
Pielou's evenness index
  Baseline: number analyzed (samples) | 45 | 42
  Baseline | 0.69 [0.25 to 0.83] | 0.69 [0.56 to 0.80]
  Post-treatment (months 1 and 6 combined): number analyzed (Participants) | 42 | 42
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 65
  Post-treatment (months 1 and 6 combined) | 0.69 [0.37 to 0.84] | 0.70 [0.45 to 0.83]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.05, Kruskal-Wallis

10. Secondary Outcome: Shannon Diversity Index of the Stool Microbiome
Description: The microbiome of study participants will be analyzed in stool samples at enrollment, week 4 and month 6 visits. Changes will be compared in the stool microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. The Shannon diversity index takes into account the number of species living in a habitat (richness) and their relative abundance (evenness). The minimum value is 0, which indicates no diversity (only one species is found). There is no upper limit to the index; the maximum value occurs when all species have the same number of individuals. Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: Shannon diversity index
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 44 | 43
Number analyzed (samples) | 113 | 111
Shannon diversity index
  Baseline: number analyzed (samples) | 44 | 43
  Baseline | 5.1 [3.5 to 6.2] | 5.3 [2.9 to 6.8]
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 68
  Post-treatment (months 1 and 6 combined) | 5.2 [3.8 to 6.3] | 5.2 [3.7 to 6.7]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.05, Kruskal-Wallis

11. Secondary Outcome: Faith's Phylogenetic Diversity of the Stool Microbiome
Description: The microbiome of study participants will be analyzed in stool samples at enrollment, week 4 and month 6 visits. Changes will be compared in the stool microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. Metagenomic analysis of deidentified selected fecal sample will be done on patients that positively respond to Theracurmin to achieve strain level identification of microbes positively and negatively associated with improved outcomes. Phylogenetic diversity (PD) is a measure of biodiversity, based on phylogeny (the tree of life). PD is defined as equal to the sum of the lengths of all the branches on the tree that span the members of the set. The branch lengths on the tree count the relative number of new features arising along that part of the tree. Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: units of PD
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 44 | 43
Number analyzed (samples) | 113 | 111
units of PD
  Baseline: number analyzed (samples) | 44 | 43
  Baseline | 10.8 [5.2 to 19.5] | 10.4 [4.8 to 17.9]
  Post-treatment (months 1 and 6 combined): number analyzed (Participants) | 40 | 38
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 68
  Post-treatment (months 1 and 6 combined) | 10.8 [4.7 to 18.1] | 10.6 [5.1 to 18.6]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.05, Kruskal-Wallis

12. Secondary Outcome: Observed Features (Amplicon Sequence Variants, ASVs) of the Stool Microbiome
Description: The microbiome of study participants will be analyzed in stool samples at enrollment, week 4 and month 6 visits. Changes will be compared in the stool microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. An amplicon sequence variant (ASV) is any one of the inferred single DNA sequences recovered from a high-throughput analysis of marker genes. Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: ASVs
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 44 | 43
Number analyzed (samples) | 116 | 111
ASVs
  Baseline: number analyzed (samples) | 44 | 43
  Baseline | 146.1 [50.0 to 268.0] | 145.7 [62.0 to 265.0]
  Post-treatment (months 1 and 6 combined): number analyzed (Participants) | 40 | 38
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 68
  Post-treatment (months 1 and 6 combined) | 148.2 [61.0 to 278.0] | 146.8 [61.0 to 272.0]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.05, Kruskal-Wallis

13. Secondary Outcome: Pielou's Evenness Index of the Stool Microbiome
Description: The microbiome of study participants will be analyzed in stool samples at enrollment, week 4 and month 6 visits. Changes will be compared in the stool microbiome over time in patients with ALS on Theracurmin to the changes observed in untreated healthy controls. Pielou's evenness is an index that measures diversity along with species richness. While species richness is the number of different species in a given area, evenness is the count of individuals of each species in an area. A calculated value of Pielou's evenness ranges from 0 (no evenness) to 1 (complete evenness). Baseline was compared to post-treatment samples from months 1 and 6 analyzed together.
Time Frame: Baseline, month 1, month 6
Population: Participants with samples collected. Post-treatment samples from months 1 and 6 were analyzed together.
Measure: Mean (Full Range); unit: Pielou's evenness index
Units Other Than Participants: samples
Arm/Group | Open Label Arm | Healthy Control Arm
Number analyzed (Participants) | 44 | 43
Number analyzed (samples) | 116 | 111
Pielou's evenness index
  Baseline: number analyzed (samples) | 44 | 43
  Baseline | 0.72 [0.55 to 0.80] | 0.74 [0.47 to 0.84]
  Post-treatment (months 1 and 6 combined): number analyzed (Participants) | 40 | 38
  Post-treatment (months 1 and 6 combined): number analyzed (samples) | 72 | 68
  Post-treatment (months 1 and 6 combined) | 0.73 [0.57 to 0.82] | 0.73 [0.56 to 0.83]
Statistical Analysis 1: Comparison: Open Label Arm; Open Label Arm participant samples from baseline, month 1, and month 6; Test type: Other; p > 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Adverse Events data not collected on the healthy control arm.
Arm/Group | Open Label Arm | Healthy Control Arm
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/0
Other Adverse Events (participants affected / at risk) | 23/50 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Arm (N=50) | Healthy Control Arm (N=0)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Arm (N=50) | Healthy Control Arm (N=0)
Diarrhea, loose stools (Gastrointestinal disorders) | 11 | 0
Hot flashes (General disorders) | 3 | 0
COVID Infection (Infections and infestations) | 3 | 0
Itching (Skin and subcutaneous tissue disorders) | 2 | 0
Increased weakness (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Flu-like symptoms (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Abdominal pain (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Cramps (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT04499963/Prot_SAP_000.pdf